CLINICAL TRIAL: NCT02731222
Title: Prevalence of Onychodystrophy in Patients With Chronic Venous Disease of the Lower Limbs
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ONI-2015-67
Record Dates: First submitted 2016-02-24; First posted 2016-04-07 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Lower Extremity Chronic Venous Insufficiency; Onychodystrophy
Keywords: CEAP classification; CVD: Chronic Venous Disease; Onychodystrophy; Body Mass Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational cross-sect. analytical inferential unicentric — collecting data from patients of the Service of Angiology and Vascular Surgery of the Hospital de Sant Pau
  Other Names: collecting data

SUMMARY:
The objective of this study is to determine the degree of correlation between the clinical severity of chronic venous disease and the prevalence of onychodystrophy. The completion of the study will require a previous synthetic explanation of the aforementioned two diseases, emphasizing the factors which have an impact on the proposed analysis.

DETAILED DESCRIPTION:
The ultimate goal of this work is to determine if patients with a higher clinical severity of chronic venous disease also present a higher prevalence of onychodystrophy. Chronic venous disease (CVD) is a vascular disease that manifests itself in the lower limbs and is related to a number of different clinical syndromes, all of which have venous hypertension (HTV) in common.

Onychodystrophy in the lower limbs is a progressive non-infectious condition associated with various factors the prevalence of which increases with age.It is mainly an acquired condition, but it can also be congenital. It is associated to a number of factors, it can sometimes be asymptomatic and it is progressive, non transmittable and evolves at a slow pace. It is characterised by an abnormal pigmentation, changes in the shape or texture and/or the deformation of nails.

The work performed was observational, cross-sectional, analytical, inferential and unicentric. In order to prove its feasibility, the researcher conducted a preliminary investigation work (pilot study) with a total of 40 patients (aged 40 to 85) who were treated at the Service of Angiology and Vascular Surgery of the Hospital de Sant Pau (Barcelona, Spain). These patients were selected to verify their data and then the researcher performed a statistical study from a descriptive and inferential point of view to find out whether there is a relation betwen the prevalence of onychodystrophy and the degree of severity of chronic venous disease. In order to minimise methodological mistakes in the outcomes and sampling, the study has been carefully defined and framed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an age ranging between 40 and 85 years.
* Patients who attend the service of Angiology, Vascular and Endovascular Surgery with chronic venous disease in their lower limbs and presenting a clinical degree according to the CEAP Classification (Clinic, Etiology, Anatomy, Pathophysiology) ranging from C0 to C6, while at the same time manifesting or not venous reflux when exposed to an echo-Doppler scan.
* Patients agreeing to voluntarily participate in the study who sign the informed consent document.

Exclusion Criteria:

* Congenital Onychopathy
* Presence in any nail plate of fungal, viral or bacterial infections
* Emergence of digital deformities in feet
* Manifestation of biomechanical problems
* Presence of advanced degenerative joint disease (arthrosis, arthritis)
* Patients who make or have made routine use of inappropriate or poorly adjusted footwear and especially those who have an onychodystrophy which is clearly and directly atributable to it
* Individuals presenting a Greek foot and especially those that present onychodystrophy on their second toe.
* Patients in which onychodystrophy is due to a surgical iatrogenic event
* Individuals with existing subungual tumours (benign or malignant).
* Patients who take or have taken any drug that causes or is directly associated with onychodystrophy
* Patients with a history of skin diseases such as psoriasis, lichen planus or alopecia areata associated with nail manifestations.
* Patients with a background of physical or chemical trauma on their toenails that has clearly given rise to onychodystrophy.
* Individuals presenting any type of amputation of the lower limbs, either in the leg or the foot, including those presenting a toe amputation (total or partial).
* Patients with a history of toenail surgery (as recent as a year or less).
* Individuals that, despite complying with all the requirements of the study, decline to participate or refuse to sign the informed consent document.
* People with any medical illness or psychiatric disorder which, in the opinion of the investigator, preclude them from understanding the reason for their selection or who were unable to give informed consent to their participation in the study.
* Subjects with post-thrombotic syndrome.
* Any affected lower limb with varicose veins having undergone surgery with any invasive procedure was excluded.
* Patients presenting nail prosthesis or cosmetics were also excluded from the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After the collection of the data, the researcher will establish the variables, including all clinical data, the Doppler echography data, the CVD symptoms, and the class to which the subject belongs according to the CEAP Classification ( ranging from 0 to 6). All these data will be analyzed in relation to the presence of onychodystrophy in each patient. Other variables that can be related to onychodystrophy will also be registered: type of footwear, feet deformation, personal history and local factors considered potentially responsible for the presence of onychodystrophy. Finally, the researcher will perform the statistical analysis relating all the variables to finally determine whether there exists or not a correlation betwen (CVD) and onychodystrophy.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2015-12-17 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
The prevalence of onychodystrophy is higher amongst patients who present a higher degree of chronic venous disease | At baseline
  The results were obtained from 83 patients, 23 men and 60 women, 40-85 years old. 120 lower limbs were analysed. All studied subjects presented CVD in the studied limb. Some presented onychodystrophy in the studied limb. Each subject was assigned a CEAP classification class (C0 to C6) depending on the severity of their CVD.
  Participants were also grouped according to age and gender to establish the relation between certain variables and the degree to which their veins are affected.
  We used descriptive and inferential statistics to estimate the population parameters, ensuring a significance level of α=0.05 to α=0.1, i. e. a degree of confidence of 90-95%. Given the statistical results and the degree of confidence, we think the main hypothesis ("The prevalence of onychodystrophy is higher amongst patients who present a higher degree of chronic venous disease") is proven and we can confirm the association between onychodystrophy in the lower limbs and CVD.

CONTACTS AND LOCATIONS:
Overall Officials: José Román Escudero, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided